CLINICAL TRIAL: NCT00034918
Title: An Open-label, Multicenter Phase II Study to Assess the Response of Subjects With Metastatic Breast Cancer Previously Treated With Anthracycline and Taxane Therapy With or Without Capecitabine to ZD6474 (100-mg or 300-mg Daily Oral Dose).
Brief Title: This Study is to Assess the Efficacy and Safety of ZD6474 in Subjects With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 6474IL/0002
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Breast Neoplasms; Metastases, Neoplasm
Keywords: Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — vandetanib

INTERVENTIONS:
Drug: ZD6474

SUMMARY:
The purpose of this study is to assess the efficacy of ZD6474 in patients with metastatic breast cancer at 2 dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Histological and/or cytological confirmation of metastatic breast cancer which is refractory to anthracycline, taxane, with or without capecitabine therapies;
* WHO performance status 0, 1 or 2 on the day of registration;
* Females, aged >= 18 years;
* No Gastrointestinal pathology which could affect the bioavailability of ZD6474.

Exclusion Criteria:

* Any evidence of severe or uncontrolled systemic diseases including known cases of Hepatitis B or C or human immunodeficiency virus (HIV).
* Significant cardiac event (including symptomatic heart failure or unstable angina) within 3 months of entry or any cardiac disease that in the opinion of the investigator increases risk for ventricular arrhythmia;
* History of clinically significant cardiac arrhythmia (multifocal PVCs, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTC grade 3) or asymptomatic sustained ventricular tachycardia;
* Chronic atrial fibrillation;
* Previous history of QT / QTc prolongation with other medication;
* Congenital long QT syndrome;
* Systemic anti-cancer therapy or other investigational agent within the last 4 weeks (6 weeks for nitrosoureas, mitomycin C, or suramin);
* Currently receiving drugs with known significant 3A4 inhibitory (ie, ketoconazole, itraconazole, troleandomycin, erythromycin, diltiazem, verapamil) or stimulatory (ie, phenytoin, carbamazepine, barbiturates, rifampicin) effects;
* Currently receiving therapeutic doses of warfarin (Coumadin?)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2002-05; Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Research Site, Indianapolis, Indiana, United States
- Research Site, Barcelona, Spain